CLINICAL TRIAL: NCT04352881
Title: Evaluation of the Management of Dental Emergencies During Night and Week-ends
Brief Title: Evaluation of Out of Hours Dental Emergency Treatments
Acronym: URGDENT-NW
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191120
Record Dates: First submitted 2020-02-26; First posted 2020-04-20 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-02

CONDITIONS: Orofacial Pain; Orofacial Edema; Dental Trauma; Oral Infection
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionary patient — Assessing pain reduction using a 4-step questionary

SUMMARY:
For 12 years, the odontology service of the Pitié-Salpêtrière hospital group (GHPS) has been responsible for day and night dental emergency care. Several surveys have been conducted in order to analyze the sociological characteristics of the patients and the typology of the acts performed. These studies indicate that pain is the main reason for consultations, cited by 60 to 80% of patients.

So far, very few studies have been done in the context of emergencies. Very recently, a study was undertaken on the satisfaction of patients consulting the odontological emergencies of the GHPS, during a thesis work.

This study, carried out in collaboration with the URC Pitié Salpêtrière, under analysis, relates to the satisfaction of patients consulting the odontological emergencies of the GHPS during the day and week, Monday to Friday, excluding night and week emergencies -end (WE).

Attendance at night and during WE is important because it is sociologically and medically different from that of day and week. It is therefore important to complete this study by focusing on patients consulting the emergency room at night and during the weekend.

This work therefore responds to a request from the Odontology Emergency Reception Service (SAUO) of the Pitié-Salpêtrière Hospital Group. It will be carried out in the form of a survey whose objective is to assess: on the one hand, the effectiveness of the care provided in this emergency functional unit, and on the other hand the satisfaction of the patients after their passage to the emergency room .

DETAILED DESCRIPTION:
I. Research progress Two investigators will take turns in the service for the search duration. They will be responsible for informing patients of the research upon their arrival in the service and for the data collection and telephone follow-ups.

The course of the research will take place as follows:

Day of consultation (D0):

1. Patient information on the search when he arrives in the service; explanation of its objectives, its modalities and constraints.
2. Verification of eligibility criteria.
3. Collection of the patient's non-opposition by the dentist during the consultation
4. Consultation according to the usual care. During this procedure, the practitioner performs a medical history and, according to the patient's answers, completes the "General Information Questionnaire".

   He carries out the emergency care and explains the postoperative consequences.
5. Patient filling in the satisfaction questionnaire immediately after consultation.

   Telephone follow-up:
6. Telephone follow-up by the interviewer and fill in the questionnaire - in case of non-availability of the patient on day 1, the patient will be recalled on day 2 and the extrapolated data on the slope of the curve between D1 and D2
7. Telephone follow-up by the interviewer on the day and filling in the questionnaire - if the patient is not available on day 3, the patient will be recalled on day 4 and the data extrapolated according to the slope of the curve between D1 and D4; if the patient is not available at D4, he will be recalled to D5 and the extrapolated data between D1 and D5.
8. Telephone follow-up on the interviewer's day and fill in the questionnaire in case of non-availability of the patient on day 7, the patient will be recalled to D8 and the data extrapolated according to the slope of the curve between D3 and D8; if the patient is still not available on D8, he will be recalled to D9 and the extrapolated data between D3 and D9.

For the night sample : from 6:30 pm to 8 am Recall should be 24 hours after the care, but it seems not ethical or efficient to recall patients the night following ; an extension of 12 hours will be instaurated, taking then the recalls to 36h (D1), 84h (D3), and 180h (D7) after the care.

For the WE sample : from 8 am to 6:30 pm D1: 24 hours after the care D3: 72 hours after the care D7 :168 hours after the care

II.1.STATISTICAL ASPECTS

II.1. Statistical justification for the sample size 58,921 patients were received in emergency consultation day and night during the year 2017. We wish to constitute a sample of 1% of the population concerned.

For the night sample The investigators are interested here in patients received in night emergencies, 26 050 patients in 2018. On average 72 patients are received daily in emergencies of day, about 504 per week.

According to a previous study in the department (15), 50% of patients in care could not be included in the study or were lost to follow-up.

This leads to a number of 252 analysable patients per week. The investigators will therefore conduct our study over 9 nights, to include 325 patients, ie 1.25% of the population consulting For the WE sample The investigators are interested here in patients received in Saturday and Sunday emergencies, 10 657 patients in 2018. On average 204 patients are received each week-end in emergencies of day.

According to a previous study in the department (15), 50% of patients in care could not be included in the study or were lost to follow-up.

This leads to a number of 102 analysable patients per week-end. The investigators will therefore conduct our study over 2 week-ends, to include 204 patients, ie 1.9% of the population consulting

II.2. Description of statistical methods A descriptive analysis of the characteristics of the sample will be performed (age, sex, reason for consultation, diagnosis, prior appointment test, average score of anxiety and pain scores on D0, D1, D3, D7, compliance with instructions and making follow-up appointments,), satisfaction rating, appreciation of the quality of medical care, politeness of staff, waiting time, assessment of the quality of the care setting, the information received, the treatment received, and the recommendation of the service to third parties will be made.

An analysis of the evolution of pain and anxiety scores between D0, D1, D3 and D7 will be performed.

Correlations between the type of treatment and the perceived pain as well as the type of treatment and the perceived anxiety will be made.

II.3. Method of taking into account missing or invalid data Patients unreachable during the telephone follow-up period will be contacted the next day; the pain and anxiety scores will then be extrapolated from the previous data and the new data collected, by calculating the nearest point on the curve connecting these two data. If they are new unreachable, the data will be considered missing. Data from patients with missing data will be analyzed separately.

III. DATA MANAGEMENT III.1. Terms of data collection The research does not foresee the use of data extracted from existing information systems or from previously completed studies.

No nominative data will be collected as part of this research. The data will be rendered non-identifying. They must not in any case show in clear the names of the persons concerned or their address.

As part of this research, topics will be identified as follows:

N or W (depending on the Night or Week-end sample) - Chronological order of the person (3 digits) - first letter of the first name - first letter of last name The answers to the different questionnaires (completed by the patients and the interviewers) will be entered into an EXCEL file. This file will be protected by a password.

The seizure will be carried out by the coordinating investigator or one of those collaborators (dentist or student) declared in the center and trained in research at the end of each session.

III.2. Data circuit The investigators will collect the data directly from the patient during the consultation or during telephone interviews on paper forms (CRF).

This data will then be entered into an Excel database specifically created for the search.

The database will be kept on the computer of the odontology service at the Pitié-Salpêtrière hospital and will be protected by a password known only to research stakeholders.

Data analysis will be done by the principal investigator and the research stakeholders

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient reachable by telephone during the week following his / her care in the service
* Collection of the consent of the patient for his participation in research
* Good understanding of the French languageExclusion Criteria:

Exclusion criteria :

-Patient with communication difficulties or difficulties in understanding the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients seeking care at the dental emergency service at night (N) or week-end (WE) (2 samples)
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Pain score evolution measured by a 0-10 numeric scale (NS) where 0 is no pain and 10 the worst pain imaginable | Day 1
  Self reported measure of pain on the numeric scale 24h (Day 1) after the first visit (Day 0)

SECONDARY OUTCOMES:
Pain score evolution measured 3 days and 7 days after 1st visit, measured with a 0-10 numeric scale (NS) where 0 is no pain and 10 the worst pain imaginable | Day 3 and Day 7
  the pain is measured with the numeric scale
welcoming quality from hospital staff | Day 1
  Perception of welcoming, waiting time will be measured with a 0-10 numeric scale where 0 is the worst score and 10 is the best score.
anxiety score | Day 0, Day 1, Day 3, Day 7
  Anxiety score evolution measured by a 0-10 numeric scale (NS) where 0 is no anxiety and 10 the worst anxiety imaginable. The patient anxiety will be measured by numeric scale at Day 0, Day+1, Day +3, Day+7
perception of the technical quality of the emergency treatment | Day 1
  The perception is measured just after care with a 0-10 NS where 0 is the worst score and 10 is the best score

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'odontologie, Hôpital Pitié-Salpêtrière, Paris, France